CLINICAL TRIAL: NCT06038929
Title: REVEAL - Research Evaluating Vagal Excitation and Anatomical Linkages Gastric Emptying Ancillary Project: Effect of Vagal Nerve Stimulation on Gastric Motor Functions
Brief Title: Effect of Vagal Nerve Stimulation on Gastric Motor Functions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Professor of Medicine, Pharmacology and Physiology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-006558
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-07

CONDITIONS: Depression; Epilepsy
MeSH Terms: conditions — Depression; Epilepsy

STUDY DESIGN:
Intervention Model Description: Single cohort, open label study in 16 Vagus Nerve Stimulant-implanted subjects with drug-resistant epilepsy with seizures or depression, aged 18 years or older
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- vagal nerve stimulant (Experimental): The aim is to measure gastric emptying and gastric accommodation in response to a caloric meal in participants who have received insertion of the VNS for the treatment of medication - resistant depression.
  Interventions: Device: Vagal nerve stimulant

INTERVENTIONS:
Device: Vagal nerve stimulant — Vagus nerve stimulation involves using a device to stimulate the vagus nerve with electrical impulses. The implanted electrodes transmit electrical impulses travel to areas of the brain to treat conditions (intractable epilepsy, depression) and also send electrical impulses to the stomach.

SUMMARY:
The specific aim of this study is to compare simultaneous assessment of gastric emptying and gastric accommodation in response to a caloric meal In patients who have previously undergone activation of left cervical VNS for the treatment of medication-resistant depression. Our hypothesis is that cervical VNS increases gastric accommodation and accelerates gastric emptying compared to a bank of healthy control data.

DETAILED DESCRIPTION:
Objectives To compare simultaneous assessment of gastric emptying and gastric accommodation in response to the same caloric meal in patients who have undergone activation of left cervical Vagal Nerve Stimulation.

Design and Outcomes Single cohort study in 12 Vagus Nerve Stimulant-implanted subjects with drug-resistant depression, aged 18 years or older who were consented for the main VESPA REVEAL Common Study Protocol.

There is only 1 visit needed, with an average time commitment of 4.5 hours. Participants will have completed their planned VESPA REVEAL study visits Interventions and Duration In this single cohort study in 12 Vagus Nerve Stimulant-implanted subjects, each participant will undergo combined gastric emptying/accommodation test after completing the Visits required in CSP

Sample Size and Population

Sample size assessment. This will be based on results of the primary endpoints in our Mayo Clinic lab. We expect 80% power, α=0.05, assuming unpaired t-test analysis with n=12 in patients receiving VNS compared to the healthy control data (n=300 for both gastric emptying and gastric volume . Demonstrable differences (Table 1) will be based on the variation (SD) observed from our Mayo Clinic prior studies.

Table 1A. Effect size demonstrable for primary endpoints of interest, based on 80% power at α=0.05 (for n=12 with p-VNS): PRIMARY ANALYSIS

Response Meal SD Effect size detectable [absolute (% of mean)]

Fasting gastric volume, mL 273 57 471mL (17.3%)

Postmeal gastric volume, mL 848 111 92mL (10.8%)

GE of solids T1/2, min 122 29.8 24.7 min (20.2%)

In addition, these effect sizes are feasible in response to vagal intervention, whether it turns out to be stimulatory or inhibitory, and a 26-minute difference in GE T1/2 is clinically significant, as documented in a published meta-regression from our research team.

Human subjects. Participants will be recruited primarily from the University of Minnesota (90-minute drive away). With only limited added burden on participants, who will previously have undergone placement of vagal nerve stimulator. There is only 1 total visits needed, with an average time commitment of 4.5 hours.

The patients will have undergone placement of the VNS for clinical indications.

The objective of the study is to evaluate the effects of this treatment on gastric functions, rather than any therapeutic intent, or the development of a new indication to be submitted to regulatory agencies for an additional therapeutic indication. Therefore, it is perceived that an application for an investigational device exemption (IDE) is not required.

ELIGIBILITY:
General criteria

1. Participant must be at least 18 years old.
2. Participant must have the capacity to provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization.
3. Participant is diagnosed with drug Resistant Epilepsy and previously underwent implantation of VNS.

   and/or
4. Participant is diagnosed with treatment-refractory depression and previously underwent implantation of VNS.
5. Participant has completed the REVEAL CSP and has been stabilized by their care team on a stable VNS setting
6. Apart from epilepsy or depression, participant should be medically and neurologically stable.
7. Participant is able to complete regular office visits and telephone appointments including the imaging session in accordance with the study protocol requirements.
8. Participant that is of childbearing potential must be adequately protected from conception or willing to use an acceptable method of birth control over the entire study duration (acceptable birth control includes abstinence, barrier methods, hormonal methods, sterilization and fertility awareness).
9. Participant must be enrolled in an active health insurance plan that will cover the costs associated with standard health care services and injuries.

Exclusion Criteria: GENERAL criteria

1. Participant has a prior implantable stimulation device other than a VNS device for the clinical indication of refractory focal Epilepsy or for depression.
2. Participant currently uses or during the study is expected to use short-wave diathermy, microwave, diathermy, or therapeutic ultrasound diathermy.
3. Participant has a diagnosis of Substance Use Disorder as defined by DSM-5 without sustained remission of 12 months or longer.
4. Patient participated in another drug or device trial within the preceding 30 days (other than REVEAL studies).
5. Participant has been hospitalized for a psychiatric condition within the preceding 6 months or has had a history of psychosis within the preceding two years (excluding post-ictal psychosis).
6. Participant has experienced unprovoked status epilepticus in the preceding year.
7. Participant is not able or willing to use their dominant arm, or either upper arm circumference is greater than 50 cm.
8. Any other clinical reasons deemed by the investigators of the study for which the participant would not be an appropriate candidate for the study, such as peripheral vascular disease, Raynaud's phenomenon, orthostatic hypotension (OH), postural orthostatic tachycardia syndrome (POTS), uncontrolled obstructive sleep apnea (OSA), chronic obstructive pulmonary disease (COPD), or uncontrolled diabetes or pregnancy
9. Participant with vocal cord paralysis
10. Participant cannot speak and read English.
11. Participant is pregnant.
12. Prohibited Therapy During Study Period: We will exclude patients on immunosuppressants, beta blockers, anticholinergics, and clonidine. Consultation with primary providers and amending some of these therapies may be allowed only if clinically indicated. In that case, participants will have to be stable on their new medication for at least one month prior to implant.
13. A body weight of over 350 pounds or 159 kilograms due to equipment limitations used in the measurements of gastric accommodation and emptying.
14. An inability to eat eggs whether due to an allergy, intolerance, or strong dislike. The gastric emptying test meal contains eggs that are labeled with radioisotope. Other food substitutions for the toast, butter and milk may be made only if prior approval is given by Dr. Camilleri.
15. Any other factor that may impact participant safety or compliance as per PI.

Since participants with pVNS will be recruited from the CSP study at U Minnesota, it is important to specify the inclusion and exclusion criteria for participants with drug-resistant epilepsy or drug-resistant depression who entered the CSP study:

Inclusion Criteria for Participants With Major Depressive Disorder That Have a Previously Implanted VNS Device

1. Participant must be at least 18 years old.
2. Participant must have the capacity to provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization.
3. Participant must be enrolled in an active health insurance plan that will cover the costs associated with standard health care services and injuries.
4. Participant must have been previously implanted with a VNS device for the clinical indication of Major Depressive Disorder (MDD).
5. Participant must have a score on the baseline administration of the Montgomery-Åsberg Depression Rating Scale (MADRS) of ≥ 22.
6. Participant must be able and willing to complete the evaluations and procedures described in the study protocol.
7. Participant must be able and willing to follow the stipulations regarding concomitant medications and excluded medications described in section 5.3 of the study protocol.
8. Participant that is of childbearing potential must be adequately protected from conception or willing to use an acceptable method of birth control over the entire study duration (acceptable birth control includes abstinence, barrier methods, hormonal methods, sterilization and fertility awareness).

Exclusion Criteria for Participants With Major Depressive Disorder That Have a Previously Implanted VNS Device

1. Participant has a prior implantable stimulation device, other than a VNS device for the clinical indication of Major Depressive Disorder (MDD).
2. Participant currently uses or is expected during the study to use short-wave diathermy, microwave, diathermy, or therapeutic ultrasound diathermy.
3. Participant is judged by the investigator to be acutely suicidal (e.g. has made specific plans or preparations to commit suicide or as indicated by the Sheehan Suicidality Tracking Scale) within the last 30 days prior to study enrollment.
4. Participant has made a suicide attempt within the previous 6 months from study enrollment.
5. Participant has a history of one or more schizophrenia-spectrum or other psychotic disorders including schizophrenia, schizoaffective disorder, delusional disorder, or a current or lifetime major depressive episode that includes psychotic features (commonly referred to as psychotic depression) according to the MINI criteria.
6. Participant has a history of significant borderline or severe personality disorder as determined by clinical judgment.
7. Participant has an active primary diagnosis of obsessive-compulsive, eating, or post-traumatic stress disorder based on the MINI criteria.
8. Participant has a diagnosis of Substance Use Disorder as defined by DSM-5 without sustained remission of 12 months or longer.
9. Participant has a presence of any type of dementia, major neurocognitive disorder, or cognitive or psychiatric deficit as determined by clinical judgment.
10. Participant has a history of rapid cycling bipolar disorder I or II.
11. Participant currently receives treatment with another investigational device or investigational drug other than the REVEAL study (or a REVEAL ancillary project or sub-study) or has participated in another drug or device trial within the preceding 30 days before enrollment.
12. Participant is not able or willing to use their dominant arm, or either upper arm circumference is greater than 50 cm.
13. Participant does not speak English.
14. Participant is pregnant.
15. Any other clinical reasons deemed by the investigators of the study for which the participant would not be an appropriate candidate for the study, such as peripheral vascular disease, Raynaud's phenomenon, orthostatic hypotension (OH), postural orthostatic tachycardia syndrome (POTS), uncontrolled obstructive sleep apnea (OSA), chronic obstructive pulmonary disease (COPD), or uncontrolled diabetes.

Inclusion Criteria for Participants With Drug Resistant Epilepsy That Have a Previously Implanted VNS Device

1. Participant must be at least 18 years old.
2. Participant must have the capacity to provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization.
3. Participant must be enrolled in an active health insurance plan that will cover the costs associated with standard health care services and injuries.
4. Participant must have been previously implanted with a VNS device for the clinical indication of drug resistant epilepsy.
5. Participant has not had demonstrable benefit from the implanted VNS device in terms of epilepsy (seizure frequency or seizure severity) or related epilepsy comorbidities (mood, cognition, quality of life), with no definite improvement or suboptimal improvement in seizure control.
6. Apart from epilepsy, the participant should be medically and neurologically stable.
7. Participant must be able and willing to complete the evaluations and procedures described in the study protocol.
8. Participant must be able and willing to follow the stipulations regarding concomitant medications and excluded medications described in section 5.3 of the study protocol.
9. Participant that is of childbearing potential must be adequately protected from conception or willing to use an acceptable method of birth control over the entire study duration (acceptable birth control includes abstinence, barrier methods, hormonal methods, sterilization and fertility awareness).

Exclusion Criteria for Participants With Drug Resistant Epilepsy That Have a Previously Implanted VNS Device

1. Participant has demonstrable benefit from implanted VNS device in terms of epilepsy (seizure frequency or seizure severity) or epilepsy comorbidity (mood, cognition, or quality of life), with seizure freedom or clinical benefit.
2. Participant has a prior implantable stimulation device, other than a VNS device for the clinical indication of refractory focal Epilepsy.
3. Participant currently uses or is expected during the study to use short-wave diathermy, microwave, diathermy, or therapeutic ultrasound diathermy.
4. Participant has been hospitalized for a psychiatric condition within the preceding 6 months or has had a history of psychosis within the preceding two years (excluding postictal psychosis).
5. Participant has experienced unprovoked status epilepticus in the preceding year.
6. Participant has a diagnosis of Substance Use Disorder as defined by DSM-5 without sustained remission of 12 months or longer.
7. Participant currently receives treatment with another investigational device or investigational drug other than the REVEAL study (or a REVEAL ancillary project or sub-study) or has participated in another drug or device trial within the preceding 30 days before enrollment.
8. Participant is not able or willing to use their dominant arm, or either upper arm circumference is greater than 50 cm.
9. Participant does not speak English.
10. Participant is pregnant.
11. Any other clinical reasons deemed by the investigators of the study for which the participant would not be an appropriate candidate for the study, such as peripheral vascular disease, Raynaud's phenomenon, orthostatic hypotension (OH), postural orthostatic tachycardia syndrome (POTS), uncontrolled obstructive sleep apnea (OSA), chronic obstructive pulmonary disease (COPD), or uncontrolled diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Gastric emptying T1/2 | during 4 hour gastric emptying test
  time to empty 50% of the whole stomach contents
Gastric accommodation | during first 1 hour of gastric emptying test
  gastric delta volume (postprandial minus fasting) for the whole stomach

SECONDARY OUTCOMES:
Gastric emptying lag time | 1 day (during gastric emptying test)
  time to empty 10% of the whole stomach
Gastric emptying 25% | 1 day (during gastric emptying test)
  time to empty 25% of the whole stomach
Gastric emptying at 2 hours | 2 hours (during gastric emptying test)
  % emptied from the whole stomach at 2h
Gastric emptying at 4 hours | 4 hours (during gastric emptying test)
  % emptied from the whole stomach at 4h
Fasting whole volume volume | baseline
  volume of whole stomach before ingestion of meal
Fasting proximal gastric volume | baseline
  volume of proximal half of stomach before ingestion of meal
Postprandial whole gastric volume | 10-30 minutes after meal ingestion
  volume of whole stomach 10-30 minutes after ingestion of meal
Postprandial proximal gastric volume | 10-30 minutes after meal ingestion
  volume of proximal half of stomach 10-30 minutes after ingestion of meal

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No